CLINICAL TRIAL: NCT07271810
Title: Association Between Primary School Children's Speaking Attitudes and Oral Health Indicators: A Cross-Sectional Study
Brief Title: Association Between Primary School Children's Speaking Attitudes and Oral Health Indicators
Status: Completed | Type: Observational
Sponsor: Ezgi Turkyilmaz (Other)
Responsible Party: Sponsor-Investigator, Ezgi Turkyilmaz, DDS, PhD - Specialist in Pediatric Dentistry, TC Erciyes University
Organization: TC Erciyes University (Other)
Other Study IDs: ERU-PEDO-2025-01; 2024/211 (Other: ERCIYES UNIVERSITY)
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Dental Caries
Keywords: Oral Health; Dental Caries; Malocclusion; Speech Attitude; Children; Primary School
MeSH Terms: conditions — Dental Caries; Malocclusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Observational Group: All participants were included in a single observational group to evaluate the relationship between speaking attitudes and oral health indicators in primary school children.
  Interventions: Other: Observational Assessment

INTERVENTIONS:
Other: Observational Assessment — This is an observational study with no intervention applied. Data were collected through clinical oral examinations and self-administered questionnaires assessing speaking attitudes and oral health-related variables.

SUMMARY:
his cross-sectional study aims to evaluate the relationship between primary school children's speaking attitudes and oral health indicators, including dental caries, malocclusion, and tooth loss. A total of 184 children aged 7-12 years participated. Sociodemographic data, oral examination findings, and Speaking Attitudes Scale for Children (SASC) scores were collected. The study seeks to identify whether oral health problems influence children's self-perceived communication confidence and to emphasize the importance of integrating oral health awareness into early educational settings.

DETAILED DESCRIPTION:
This cross-sectional observational study was conducted to assess the association between primary school children's speaking attitudes and their oral health status. The study included 184 children aged 7-12 years who underwent intraoral examinations to record dental caries (dmft/DMFT indices), malocclusion, and tooth loss. The Speaking Attitudes Scale for Children (SASC) was used to evaluate children's attitudes toward their speaking skills. Data were analyzed to explore correlations between SASC scores and oral health indicators. The findings are expected to provide insight into how oral health conditions, such as untreated caries or malocclusion, may influence children's communication confidence and social participation. Ethical approval for this study was obtained from the Erciyes University Clinical Research Ethics Committee (Approval No: 2024/211).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7-12 years enrolled in primary schools Children who are native Turkish speakers Children without systemic or developmental disorders Children and parents who provided informed consent to participate

Exclusion Criteria:

* hildren with speech or hearing impairments Children with fixed orthodontic appliances Children with missing permanent first molars due to extraction Children with a history of craniofacial anomalies or trauma

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study included 184 primary school children aged 7 to 12 years who were attending public schools in Turkey. Both male and female children were included. Participants represented a generally healthy pediatric population without chronic medical conditions.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Association between speaking attitude scores and oral health indicators | Single assessment at baseline (cross-sectional study)
ssociation between speaking attitude scores and oral health indicators | Single assessment at baseline (cross-sectional study)
  The primary outcome was the relationship between speaking attitude scores (measured by the Speaking Attitude Scale for Primary School Children) and oral health indicators such as dental caries experience (DMFT/dmft), malocclusion, and tooth loss. Higher speaking attitude scores indicate more positive speaking attitudes.
Association between speaking attitude scores and oral health indicators | Single assessment at baseline (cross-sectional study)
  The primary outcome was the relationship between speaking attitude scores (measured by the Speaking Attitude Scale for Primary School Children) and oral health indicators such as dental caries experience (DMFT/dmft), malocclusion, and tooth loss. Higher speaking attitude scores indicate more positive speaking attitudes.

SECONDARY OUTCOMES:
Relationship between oral health status and sociodemographic factors | Single assessment at baseline
  Secondary analysis included evaluating the association between children's oral health indicators (DMFT/dmft, malocclusion, tooth loss) and sociodemographic factors such as age, gender, and parental education level.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)